CLINICAL TRIAL: NCT06075992
Title: Investigation of the Effect of Infant Massage Applied in the Intensive Care Unit on Motor Performance and Stress Hormones in Premature Infants
Brief Title: Massage Application and Motor Performance, Stress Assessment in Premature Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Gulsun Ceren Yalcin, Principal Investigator, Mustafa Kemal University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: fzt.cerenyalcin2023
Record Dates: First submitted 2022-12-29; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Infant; Premature Birth
Keywords: Premature baby; Newborn intensive care; Baby massage; Cortisol hormone; Motor development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premature babies in this group will be massaged. (Experimental): On the first day of the study and at the end of the 4th week, the Infant Motor Performance Test (TIMP) will be used to evaluate the infant's motor performance consisting of postural control and selective extremity movements. Anthropometric measurements of all babies included in the study immediately afterwards; The baby's body weight, height and head circumference will be checked on the first day of the study and at the end of the 4th week. The stress level of babies will be evaluated by looking at cortisol and ACTH (Adrenocorticotropic hormone) hormones. Massage therapy will be given according to the Field medium pressure massage therapy protocol. In addition to the medical treatment, the application group will be massaged by an experienced physiotherapist according to the Field baby massage therapy protocol, at least 1 hour after the babies are fed, 3 days a week, 2 times a day and for 4 weeks.The massage will be applied for 15 minutes.
  Interventions: Other: experimental group
- An experimental application will not be made to premature babies in this group. (No Intervention): No application will be made other than medical treatment. On the first day of the study and at the end of the 4th week, the Infant Motor Performance Test (TIMP) will be used to evaluate the infant's motor performance consisting of postural control and selective extremity movements. Anthropometric measurements of all babies included in the study immediately afterwards; The baby's body weight, height and head circumference will be checked on the first day of the study and at the end of the 4th week. The stress level of babies will be evaluated by looking at cortisol and ACTH (Adrenocorticotropic hormone) hormones.

INTERVENTIONS:
Other: experimental group — An experimental application will not be made to premature babies in this group.
  Other Names: No Intervention group
  Arms: Premature babies in this group will be massaged.

SUMMARY:
In our study, the effect of infant massage applied in the intensive care unit on motor performance and stress hormones in premature babies will be examined. The number of patients to participate in the study was determined as 30. Appropriate babies will be determined and divided into 2 groups by drawing lots. After recording the demographic information of the babies who meet the inclusion criteria, the Baby Motor Performance Test (TIMP) and the baby's motor performance evaluation consisting of postural control and selective extremity movements, and the stress level of the babies will be evaluated by looking at cortisol and adrenocorticotropic hormone (ACTH) hormones. In addition, Field baby massage will be given to the application group. It is seen that there are limited studies in the literature on the effect of infant massage applied in the intensive care unit on motor performance and stress hormones in premature infants. The results of this research will provide useful information for premature babies hospitalized in intensive care.

DETAILED DESCRIPTION:
The time a baby spends in the womb is gestational age. This period can vary between 37 and 42 weeks. gestational week (GH); It is the number of weeks from the mother's last menstrual cycle to the birth of the baby. Term birth is considered as the birth that occurs after the completion of this period. The first 28-day period after birth is called the "newborn period" . Premature birth is defined as live births that occur before 37 weeks of gestation are completed. According to the data of the World Health Organization (WHO); About 15 million premature babies are born in the world every year. It is known that 1 million of the babies born died only due to complications related to premature birth. While the rate of preterm birth varies between 5% and 18% in the world, this rate is estimated to be between 10% and 15% for Turkey. Although prematurity is the most important cause of neonatal mortality and morbidity, it is reported to be responsible for 40% of deaths under 5 years of age. In the studies carried out; It has been found that the risk of developing sequelae is significantly higher in babies born before the 33rd week of birth and classified as very premature babies and extremely premature babies, compared to late premature babies and term babies, since their brain development is not completed.

Neonatal intensive care unit (NICU); health care provider is considered as part of perinatal care. In addition, they are units that serve term and premature babies who need high quality medical and surgical treatments. When the premature baby is in a critical period for brain development, he is separated from the warm, dark, quiet mother's womb, which is suitable for brain development, and placed in a loud, bright light, crowded and complex NICU. It is also full of painful medical procedures performed by connecting the premature baby to various devices such as vascular access, nasogastric and endotracheal tubes in the NICU. From the first moment of life, infants hospitalized in the NICU are frequently exposed to these stressors. Especially in premature babies, the effects of these stressors are high. Appropriate interventions are needed to improve autonomic nervous system performance because premature babies cannot fully adapt to environmental stress factors in the NICU.

Supportive care practices can be used as an approach to accelerate the development of infants and reduce complications caused by prematurity. The majority of research over the past three decades has focused on different approaches to reducing stress in infants in the NICU. These approaches are; visual, auditory and tactile stimuli, family-centered care, kangaroo care (skin to skin contact), music concert, breastfeeding support system, oral stimulation and baby massage. The aim of all these techniques is to improve the quality of life of premature babies, and it has been reported that the applications are highly effective. Massage can be defined as "a methodological touch aimed at stimulating the baby". Massage therapy can be applied using various techniques. It is the systematic application of tactile stimulation that results in the stimulation of sensory receptors in the skin, muscles, bones and joints. The mechanism of action in the infant is thought to be related to an effect on the neuroendocrine stress response system as a result of stimulation of the vagal nerve through the activation of pressure receptors. Many studies have shown the positive effects of massage therapy in preterm babies. These positive effects include weight gain, reduction in stress levels, improvement in sleep or wakefulness, early discharge from the NICU, improvement in skin integrity, increased development of the sympathetic nervous system, and increased parent-infant bond. Massage can be applied easily by families, and it can also be frequently preferred by many families to improve infant health and facilitate parent-infant bonding. In addition, it has been shown that there is strong evidence that infant massage has positive effects for infants and their parents, and reduces pain during painful procedures such as heel stick and tape removal. Although a great deal of research has been done on infant massage in NICU, the available literature is limited due to significant differences between studies in terms of massage techniques used and measured results. Various massage techniques have been used, but the most studied massage technique was developed by Field (1986). It has been suggested that when the Field protocol is applied appropriately in the form of 15-minute medium-pressure systematic tactile and kinesthetic stimulation, it can reduce stress and improve the developmental outcomes of the baby. This protocol was chosen because it has been shown that at least 15 minutes of tactile and kinesthetic intervention has beneficial effects on growth and motor activity in preterm infants. In 2006, the American Academy of Pediatrics published guidelines for the follow-up of premature babies. According to the guidelines; It has been stated that all very low birth weight and preterm infants should undergo age-appropriate motor assessment at least twice in the first year of life.

Evaluation of premature babies in the earliest period; It is important in terms of determining the appropriate treatment options for their needs and determining the early rehabilitation program.

Infant Motor Performance Test (TIMP) is a functional motor skill test with age standards for the performance of infants from the 34th week postmenstrual to the 17th postnatal week. TIMP has ecological validity to capture the infant's ability to respond to movements that reflect daily life interactions with parents during activities such as bathing, dressing, and playing. TIMP can catch the delay regardless of the underlying cause. It has been shown to be effective in educating parents about motor development in preterm infants, useful for planning intervention and evaluating treatment outcomes, and being a powerful outcome assessment tool for use in clinical studies. It has also been proven to have an important ability to predict long-term motor and cognitive outcomes. Studies on massage have reported many beneficial effects in preterm infants, including lower serum cortisol levels, increased short-term weight gain, and reduced stress with a shorter hospital stay. Cortisol is the most commonly used biochemical measurement of stress hormones, which occurs as a result of physiological changes caused by stress in newborn babies. Cortisol is defined as a "biological marker of psychological stress". ACTH (Adrenocorticotropic hormone) is a hormone that stimulates the production of cortisol. Stress stimulates ACTH production in the pituitary gland. In response, there is an increase in glucocorticoid hormone secretion by the adrenal cortex. One of these glucocorticoid hormones is cortisol, which can serve as an indicator of stress. It has been scientifically proven that massage reduces both cortisol and norepinephrine levels and causes relaxation by further increasing vagal tone. One study showed that preterm infants who received Field massage had lower amounts of urinary cortisol than those who were not treated with massage. The aim of our study is to examine the effect of infant massage applied in the intensive care unit on motor performance and stress hormones in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* 28.-34. Premature infants with stable clinical conditions born between gestational weeks,
* Babies of families whose parents can speak and understand Turkish at least one of their parents,
* Body weight over 1000 g,
* Premature babies are only due to non-invasive intubation,
* Stability of the baby's vital signs
* The baby does not have a chest tube.

Exclusion Criteria:

* Babies whose family consent cannot be obtained,
* Babies born from triplet or more multiple pregnancies,
* Babies using antiepileptic drugs,
* Medically unstable infants,
* Having a major anomaly,
* Having undergone a surgical procedure.

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline cortisol and ACTH (Adrenocorticotropic hormone) hormones at 4 weeks. | baseline and after 4 weeks
  The stress level will be evaluated by looking at the cortisol and ACTH (Adrenocorticotropic hormone) hormones of the babies.
  Infants admitted to the NICU will have their blood values routinely checked at regular intervals by the infant's responsible physician. The blood taken for the study will be centrifuged in a gel-free biochemistry tube.
Change from Baseline Test of Infant Motor Performance-TIMP at 4 weeks. | baseline and after 4 weeks
  TIMP is a test battery developed for the evaluation of selective and postural control in early infancy. The Infant Motor Performance Test (TIMP) is the only differential assessment and prognosis tool developed for preterm infants of 34 weeks to 4 months of corrected gestational age with a high predictive value for use in the neonatal unit. This test is a test that evaluates motor performance, postural and selective motor control of newborns at risk of motor delay. TIMP, which was developed for the use of physiotherapists, has Turkish reliability and validity. The test begins with a 2-3 minute observation of spontaneous movement of the baby in the supine position. The first part consists of 13 items and evaluates the observational spontaneous motor movements of the baby. Items based on observation are evaluated with two options. The second part is; It consists of 29 items and a total of 42 items based on the baby's performance.
Change from Baseline height measurements at 4 weeks. | baseline and after 4 weeks
  Height measurements will be measured in centimeters. In the study, the height measurements of the babies will be made by the researcher using a non-flexible tape measure in the NICU in accordance with the measurement technique. The difference between the baby's first and second measurements will be calculated. It will be compared with the control group.
Change from Baseline head circumference measurements at 4 weeks. | baseline and after 4 weeks
  Head circumference measurements will be measured in centimeters. In the study, the head circumference measurements of the babies will be made by the researcher using a non-flexible tape measure in the NICU in accordance with the measurement technique. The difference between the baby's first and second measurements will be calculated. It will be compared with the control group.
Change from Baseline body weight at 4 weeks. | baseline and after 4 weeks
  Body weight will be measured in kilograms. body weight of the premature baby will be measured by the researcher. The measurement will be made with babies naked, wearing clean cloths. After the measurement, the actual weight of the baby will be recorded by subtracting the weight of the diaper from the body weight of the baby. The difference between the baby's first and second measurements will be calculated. It will be compared with the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha bezgin, Study Director — Hatay Mustafa Kemal University, Faculty of Health Sciences
Locations (2):
- Turkey (Türkiye) (2):
  - Hatay Mustafa Kemal University, Hatay, Antakya
  - Mustafa Kemal University, Hatay, Antakya

IPD SHARING:
Plan to Share IPD: No
As the work has not started yet, a decision has not been made.